CLINICAL TRIAL: NCT03901534
Title: Assessment of Continuous Positive Airway Pressure Therapy in OSA and ILD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanja Jelic, Associate Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6902; 1R01HL137234-01 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Interstitial Lung Disease; Obstructive Sleep Apnea
Keywords: Interstitial Lung Disease (ILD); Obstructive Sleep Apnea (OSA); CPAP
MeSH Terms: conditions — Lung Diseases, Interstitial; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Community based Multi-Ethnic Study of Atherosclerosis (MESA) (No Intervention): This cohort includes biospecimens collected from 1852 participants in the MESA sleep study [Chen et al]. Serum biomarkers were measured by immunoassay in the Laboratory for Clinical Biochemistry Research at the University of Vermont.
  All participants in this cohort will be analyzed for only the Aim 1 outcome measures.
- HeartBEAT and BestAir (No Intervention): The cohort includes 62 men and 20 women with newly diagnosed moderate-to-severe OSA and without known severe lung disease, who had participated in either of two randomized trials of PAP therapy, the HeartBEAT [Gottlieb et al] and BestAIR [Bakker et al] studies. Participants were selected for this analysis based on mean PAP adherence of ≥4 hours daily over a follow-up period of 3 months in the HeartBEAT study and 6 months in the BestAIR study.
  Morning serum samples drawn at baseline and at the end of the PAP treatment period were assayed using commercially available ELISA for each biomarker in the Laboratory for Clinical Biochemistry Research at the University of Vermont Larner College of Medicine.
  All participants in this cohort will be analyzed for only the Aim 2 outcome measures.
- CPAP treatment of OSA (Experimental): Participants with obstructive sleep apnea (OSA) will be treated with continuous positive airway pressure therapy (CPAP).
  All participants in this cohort will be analyzed for only the Aim 3a outcome measures.
  Interventions: Device: Continuous positive airway pressure (CPAP) therapy
- ILD screening for OSA (Experimental): Participants with interstitial lung disease (ILD) will be screened for OSA by polysomnography.
  All participants in this cohort will be analyzed for only the Aim 3b outcome measures.
  Interventions: Device: Nox A1 Recorder

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) therapy — Standard, clinically used CPAP therapy. CPAP will be prescribed by the participants' clinician provider and not by the study investigators.
  Arms: CPAP treatment of OSA
Device: Nox A1 Recorder — Non-invasive, body-worn, sleep recording device for nocturnal polysomnography.
  Arms: ILD screening for OSA

SUMMARY:
The purpose of this study is to evaluate whether biomarkers of lung epithelial and endothelial injury are associated with obstructive sleep apnea (OSA) and interstitial lung disease (ILD).

DETAILED DESCRIPTION:
This study is comprised of 3 aims:

Aim 1: Determine whether the greater OSA severity is associated with higher levels of serum biomarkers of AEC and endothelial injury and ECM remodeling in community-dwelling adults. This is a retrospective study that will analyze biospecimens from those who participated in the MESA sleep study [Chen et al].

Aim 2: Determine whether CPAP use is associated with reductions in alveolar epithelial cell (AEC) injury and endothelial injury, and extracellular matrix (ECM) remodeling biomarkers in adults with moderate-to-severe OSA. This is a retrospective study that will analyze biospecimens from those who participated in either the HeartBEAT [Gottlieb et al] and BestAIR [Bakker et al] studies.

Revised Aim 3: a) Determine whether untreated OSA promotes AEC and endothelial injury and ECM remodeling biomarkers in adults with ILD and OSA compared with those without OSA; b) Determine prospectively whether clinically-initiated 4-week PAP therapy increases markers of alveolar endothelial lung injury in OSA. Participants will be recruited at Columbia University and be assigned CPAP therapy as an intervention.

ELIGIBILITY:
Inclusion Criteria for Patients with ILD:

1. Ability to provide informed consent.
2. Age 18 years or greater
3. Diagnosis of any of the following fibrotic interstitial lung diseases as defined by ATS/ERS/JRS/ALAT guidelines and research statements and Delphi surveys:

   * Idiopathic pulmonary fibrosis
   * Idiopathic non-specific interstitial pneumonia (NSIP) with fibrosis
   * Chronic hypersensitivity pneumonitis with fibrosis
   * Connective tissue disease related interstitial lung disease (CTD-ILD)
   * Unclassifiable idiopathic interstitial pneumonia with fibrosis

Exclusion criteria for Patients with ILD:

1. Clinically significant lung disease other than fibrotic interstitial lung disease
2. Planned change to the IPF treatment during the study period
3. Current cigarette smoking (past 4 weeks)
4. Lower respiratory tract infection in past 60 days. (Upper respiratory tract infection is not a contraindication)
5. History of life-threatening cardiac arrhythmias
6. Known chronic heart failure (LVEF < 45% or echo evidence of RV dysfunction or PH)
7. Chronic opiate analgesic use
8. History of sleepiness-related automobile accident within past year of enrollment
9. Expected survival time in the opinion of the investigator of less than 6 months
10. History of stroke or spinal cord injury

Inclusion criteria for OSA patients:

1. Age 18 years or greater
2. Clinical diagnosis of untreated OSA documented by nocturnal polysomnography

Exclusion criteria for OSA patients:

1. Current treatment with CPAP or oral appliance
2. Identical exclusion criteria as for ILD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2021 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Researchers will be required to submit a written request to the Study Principal Investigator (PI) describing the use of the specimens. The researcher must also document institutional review board (IRB) approval and sign a material transfer agreement. The Study PI will make all decisions about use of the specimens. No identifiable information will be released, only coded anonymized samples and non-identifiable clinical/demographic information. For genomic data generated from whole-exome sequencing, the genotype and relevant phenotype data for participants who consented to share data will be registered and shared through the database of Genotypes and Phenotypes (dbGaP), a controlled access database, once the sequencing data have been cleaned and quality control procedures are completed.
Supporting Information: Study Protocol
Time Frame: Data will be available no later than 3 years after last research subject is enrolled in the study.
Access Criteria: Researchers will be required to submit a written request to the Study PI describing the use of the specimens. The researcher must also document IRB approval and sign a material transfer agreement. The Study PI will make all decisions about use of the specimens. No identifiable information will be released, only coded samples and non-identifiable clinical/demographic information.

REFERENCES:
- [Background] Chen X, Wang R, Zee P, Lutsey PL, Javaheri S, Alcantara C, Jackson CL, Williams MA, Redline S. Racial/Ethnic Differences in Sleep Disturbances: The Multi-Ethnic Study of Atherosclerosis (MESA). Sleep. 2015 Jun 1;38(6):877-88. doi: 10.5665/sleep.4732. PMID 25409106
- [Background] Gottlieb DJ, Punjabi NM, Mehra R, Patel SR, Quan SF, Babineau DC, Tracy RP, Rueschman M, Blumenthal RS, Lewis EF, Bhatt DL, Redline S. CPAP versus oxygen in obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2276-85. doi: 10.1056/NEJMoa1306766. PMID 24918372
- [Background] Bakker JP, Wang R, Weng J, Aloia MS, Toth C, Morrical MG, Gleason KJ, Rueschman M, Dorsey C, Patel SR, Ware JH, Mittleman MA, Redline S. Motivational Enhancement for Increasing Adherence to CPAP: A Randomized Controlled Trial. Chest. 2016 Aug;150(2):337-45. doi: 10.1016/j.chest.2016.03.019. Epub 2016 Mar 24. PMID 27018174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for Aim 3b of the study was terminated before any prospective participants could be enrolled.
Groups:
- Community Based Multi-Ethnic Study of Atherosclerosis (MESA): This cohort includes biospecimens collected from 1852 participants in the MESA sleep study [Chen et al]. Serum biomarkers were measured by immunoassay in the Laboratory for Clinical Biochemistry Research at the University of Vermont.
- HeartBEAT and BestAir: This cohort includes 62 men and 20 women with newly diagnosed moderate-to-severe OSA and without known severe lung disease, who had participated in either of two randomized trials of PAP therapy, the HeartBEAT [Gottlieb et al] and BestAIR [Bakker et al] studies. Participants were selected for this analysis based on mean PAP adherence of =4 hours daily over a follow-up period of 3 months in the HeartBEAT study and 6 months in the BestAIR study.
  Morning serum samples drawn at baseline and at the end of the PAP treatment period were assayed using commercially available ELISA for each biomarker in the Laboratory for Clinical Biochemistry Research at the University of Vermont Larner College of Medicine.
- CPAP Treatment of OSA: Participants with obstructive sleep apnea (OSA) will be treated with continuous positive airway pressure therapy (CPAP).
- ILD Screening for OSA: Participants with interstitial lung disease (ILD) will be screened for OSA by polysomnography.
Period: Aim 1
Arm/Group | Community Based Multi-Ethnic Study of Atherosclerosis (MESA) | HeartBEAT and BestAir | CPAP Treatment of OSA | ILD Screening for OSA
Started | 1852 | 0 | 0 | 0
Completed | 1852 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Aim 2
Arm/Group | Community Based Multi-Ethnic Study of Atherosclerosis (MESA) | HeartBEAT and BestAir | CPAP Treatment of OSA | ILD Screening for OSA
Started | 0 | 82 | 0 | 0
Completed | 0 | 82 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Aim 3a
Arm/Group | Community Based Multi-Ethnic Study of Atherosclerosis (MESA) | HeartBEAT and BestAir | CPAP Treatment of OSA | ILD Screening for OSA
Started | 0 | 0 | 87 | 0
Completed | 0 | 0 | 87 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Aim 3b
Arm/Group | Community Based Multi-Ethnic Study of Atherosclerosis (MESA) | HeartBEAT and BestAir | CPAP Treatment of OSA | ILD Screening for OSA
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled for Aim 3b.
Groups:
- Aim 1 Cohort: MESA: This cohort includes biospecimens collected from 1852 participants in the MESA sleep study [Chen et al]. Serum biomarkers were measured by immunoassay in the Laboratory for Clinical Biochemistry Research at the University of Vermont.
- Aim 2 Cohort: HeartBEAT and BestAir: This cohort includes 62 men and 20 women with newly diagnosed moderate-to-severe OSA and without known severe lung disease, who had participated in either of two randomized trials of PAP therapy, the HeartBEAT [Gottlieb et al] and BestAIR [Bakker et al] studies. Participants were selected for this analysis based on mean PAP adherence of =4 hours daily over a follow-up period of 3 months in the HeartBEAT study and 6 months in the BestAIR study.
  Morning serum samples drawn at baseline and at the end of the PAP treatment period were assayed using commercially available ELISA for each biomarker in the Laboratory for Clinical Biochemistry Research at the University of Vermont Larner College of Medicine.
- Aim 3a Cohort: CPAP Treatment of OSA: Participants with OSA will be treated with CPAP.
- Aim 3b Cohort: ILD Screening for OSA: Participants with ILD will be screened for OSA by polysomnography.
- Total: Total of all reporting groups
Arm/Group | Aim 1 Cohort: MESA | Aim 2 Cohort: HeartBEAT and BestAir | Aim 3a Cohort: CPAP Treatment of OSA | Aim 3b Cohort: ILD Screening for OSA | Total
Number analyzed (Participants) | 1852 | 82 | 87 | 0 | 2021
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9) | 65 (7) | 46 (13) |  | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 979 | 20 | 41 |  | 1040
  Male | 873 | 62 | 46 |  | 981
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1852 | 82 | 87 |  | 2021

OUTCOME MEASURES:

1. Primary Outcome: Surfactant Protein D (SP-D) [Aim 1]
Description: SP-D is a marker of alveolar epithelial cell injury.
  This Outcome is specific to Aim 1 and will only be measured on participants in the Aim 1 phase of the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- MESA: This cohort includes biospecimens collected from 1852 participants in the MESA sleep study [Chen et al]. Serum biomarkers were measured by immunoassay in the Laboratory for Clinical Biochemistry Research at the University of Vermont.
Arm/Group | MESA
Number analyzed (Participants) | 1852
pg/mL | 8 (6)

2. Primary Outcome: E-selectin [Aim 1]
Description: This Outcome is specific to Aim 1 and will only be measured on participants in the Aim 1 phase of the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MESA
Number analyzed (Participants) | 1852
pg/mL | 20438 (10558)

3. Primary Outcome: Angiopoietin-2 [Aim 1]
Description: This Outcome is specific to Aim 1 and will only be measured on participants in the Aim 1 phase of the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MESA
Number analyzed (Participants) | 1852
pg/mL | 1785 (1082)

4. Primary Outcome: Vascular Endothelial Growth Factor-A (VEGF-A) [Aim 1]
Description: This Outcome is specific to Aim 1 and will only be measured on participants in the Aim 1 phase of the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MESA
Number analyzed (Participants) | 1852
pg/mL | 156 (125)

5. Primary Outcome: Angiopoietin-interacting Soluble Tie-2 (sTie2) [Aim 1]
Description: This Outcome is specific to Aim 1 and will only be measured on participants in the Aim 1 phase of the study.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MESA
Number analyzed (Participants) | 1852
pg/mL | 83496 (15417)

6. Primary Outcome: Change in Serum Matrix Metalloproteinase-7 (MMP-7) Following CPAP [Aim 2]
Description: The differences between-arms in the longitudinal changes of MMP-7 will be measured. For the purpose of this analysis, all individuals receiving active CPAP in the experimental arm will be compared to all individuals receiving sham CPAP device in the control arm.
  This Outcome is specific to Aim 2 and will only be measured on participants in the Aim 2 phase of the study.
Time Frame: Baseline and post-CPAP follow-up, up to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- HeartBEAT and BestAir: This cohort includes 62 men and 20 women with newly diagnosed moderate-to-severe OSA and without known severe lung disease, who had participated in either of two randomized trials of PAP therapy, the HeartBEAT [Gottlieb et al] and BestAIR [Bakker et al] studies. Participants were selected for this analysis based on mean PAP adherence of ≥4 hours daily over a follow-up period of 3 months in the HeartBEAT study and 6 months in the BestAIR study.
  Morning serum samples drawn at baseline and at the end of the PAP treatment period were assayed using commercially available ELISA for each biomarker in the Laboratory for Clinical Biochemistry Research at the University of Vermont Larner College of Medicine.
Arm/Group | HeartBEAT and BestAir
Number analyzed (Participants) | 82
ng/mL | 0.004 [-0.25 to 0.26]

7. Primary Outcome: Change in Serum Surfactant Protein-D (SP-D) Following CPAP [Aim 2]
Description: The between-arm difference in the longitudinal changes of SP-D will be measured. For the purpose of this analysis, all individuals receiving active CPAP in the experimental arm will be compared to all individuals receiving sham CPAP device in the control arm.
  This Outcome is specific to Aim 2 and will only be measured on participants in the Aim 2 phase of the study.
Time Frame: Baseline and post-CPAP follow-up, up to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HeartBEAT and BestAir
Number analyzed (Participants) | 82
ng/mL | 0.68 [-0.18 to 1.53]

8. Primary Outcome: Change in Serum Angiopoietin-2 (Ang-2) Following CPAP [Aim 2]
Description: The between-arm difference in the longitudinal changes of Ang-2 will be measured. For the purpose of this analysis, all individuals receiving active CPAP in the experimental arm will be compared to all individuals receiving sham CPAP device in the control arm.
  This Outcome is specific to Aim 2 and will only be measured on participants in the Aim 2 phase of the study.
Time Frame: Baseline and post-CPAP follow-up, up to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HeartBEAT and BestAir
Number analyzed (Participants) | 82
ng/mL | 0.28 [0.08 to 0.48]

9. Primary Outcome: Change in Serum Osteopontin Following CPAP [Aim 2]
Description: The differences between-arms in the longitudinal changes of Osteopontin will be measured. For the purpose of this analysis, all individuals receiving active CPAP in the experimental arm will be compared to all individuals receiving sham CPAP device in the control arm.
  This Outcome is specific to Aim 2 and will only be measured on participants in the Aim 2 phase of the study.
Time Frame: Baseline and post-CPAP follow-up, up to 24 Weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | HeartBEAT and BestAir
Number analyzed (Participants) | 82
ng/mL | -0.80 [-5.97 to 4.36]

10. Primary Outcome: Serum Angiopoietin-2 (Ang-2, ng/mL) [Aim 3a]
Description: Participants will be treated with CPAP for 4 weeks. Serum Ang-2 levels will be measured at baseline and after CPAP therapy.
  This Outcome is specific to Aim 3a and will only be measured on participants in the Aim 3a phase of the study.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- CPAP Treatment of OSA: Participants with OSA will be treated with CPAP.
Arm/Group | CPAP Treatment of OSA
Number analyzed (Participants) | 87
pg/mL
  Baseline | 1889 (903)
  4 weeks | 2153 (926)

11. Other Pre Specified Outcome: Serum Surfactant Protein-A (SP-A, ng/mL)
Description: The between-arm difference in the longitudinal changes of SP-A will be measured.
Time Frame: Up to 24 weeks
Population: Data was not collected thus cannot be analyzed.
Arm/Group | MESA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Adverse events were not collected from the Aim 3b cohort due to early study termination.
Arm/Group | Aim 1 Cohort: MESA | Aim 2 Cohort: HeartBEAT and BestAir | Aim 3a Cohort: CPAP Treatment of OSA | Aim 3b Cohort: ILD Screening for OSA
All-Cause Mortality (participants affected / at risk) | 0/1852 | 0/82 | 0/87 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1852 | 0/82 | 0/87 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1852 | 0/82 | 0/87 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT03901534/Prot_SAP_000.pdf